CLINICAL TRIAL: NCT04716218
Title: Effect of Back up Head Elevated Position on Laryngeal Visualization With the Video-laryngoscope in Patients With Simulated Difficult Airway.
Brief Title: Effect of Back up Head Elevated Position on Laryngeal Visualization.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jun joohyun, Associate professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-09-009
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neutral position (Placebo Comparator): The initial percentage of glottic opening (POGO) by laryngoscopy was recorded in the ramped position. Thereafter, a second POGO (laryngeal view) was scored in the neutral position and then intubation was performed.
  Interventions: Procedure: back up head elevated position
- back up head elevated position (Experimental): The initial POGO was recorded in the neutral position. The second POGO was scored in the ramped position and then the trachea was intubated.
  Interventions: Procedure: back up head elevated position

INTERVENTIONS:
Procedure: back up head elevated position — The patient was then placed in the back-up position to align the external auditory meatus and sternal notch, which was achieved by breaking the operating table at the hips to prevent patients from sliding off the table.

SUMMARY:
In patients with limited neck extension and mouth opening due to reasons including previous radiation therapy in the head and neck area or cervical spine pathology, tracheal intubation with direct laryngoscopy (DL) are challenging because of the difficulty in aligning the oral, pharyngeal, and laryngeal axes in order to visualize the cords. In contrast, video-laryngoscopes (VL) only require alignment of the pharyngeal and laryngeal axes, which lie along much more similar angles when compared with the oral axis. Thus, VL make tracheal intubation easier to accomplish in these patients.

Good patient positioning also maximizes the chance of successful laryngoscopy and tracheal intubation. In difficult airway society 2015 guidelines, advantages of head-up positioning and ramping, which brings the patient's sternum onto the horizontal plane of the external auditory meatus (EAM), are highlighted. In the obese patient, the 'ramped' position should be used routinely because this improves the view during DL. This position is usually achieved by placing blankets or other devices under the patient's head and shoulders, but can also be achieved simply by configuring the operation room (OR) table into a back-up head elevated (BUHE) position. Significantly improved glottic views on DL have been reported with both obese and non-obese adult patients in BUHE position. However, the effect of this simple maneuver on laryngeal visualization with the VL in patients with limited neck extension and mouth opening has not been reported.

The investigators hypothesized that BUHE position might improve laryngeal views and make intubation easier compared to the supine position with the VL in patients with simulated difficult airway (application of a cervical collar to limit mouth opening and neck movement).The investigator investigated primarily the improvement in visualization of the glottis and, secondarily, the ease of tracheal intubation after alignment of the EAM and sternal notch.

ELIGIBILITY:
Inclusion Criteria:

* patients of ASA physical status 1-2 who were scheduled for elective surgery under general anaesthesia requiring tracheal intubation

Exclusion Criteria:

* if they required rapid sequence induction; had a history of previous difficult direct laryngoscopy and required awake tracheal intubation; were unable or unwilling to provide informed consent; had uncontrolled hypertension; had a history of ischaemic heart disease without optimal control of symptoms; had a history of acute or recent stroke or myocardial infarction; had cervical spine instability or cervical myelopathy; had symptomatic asthma or reactive airway disease requiring daily pharmacological treatment for control of symptoms; or had a history of gastric reflux.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
POGO score | During laryngeal visualization by laryngoscope over 1 minute period
  percentage of glottic opening

SECONDARY OUTCOMES:
intubation time | The time from the insertion of laryngoscope into oral cavity until its removal over 1 minute period
  time required for intubation
ease of tracheal intubation | The time from the insertion of laryngoscope into oral cavity until tracheal intubation over 1minute period
  number of optimization procedure to facilitate laryngeal visualization and tracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chun EH, Chung MH, Kim JE, Kim KM, Lee HS, Son JM, Park J, Jun JH. Effects of head-elevated position on tracheal intubation using a McGrath MAC videolaryngoscope in patients with a simulated difficult airway: a prospective randomized crossover study. BMC Anesthesiol. 2022 May 30;22(1):166. doi: 10.1186/s12871-022-01706-5. PMID 35637437